CLINICAL TRIAL: NCT02732119
Title: A Phase I/II, Single Arm, Open-label Study of Ribociclib in Combination With Everolimus + Exemestane in the Treatment of Men and Postmenopausal Women With HR+, HER2- Locally Advanced or Metastatic Breast Cancer Following Progression on a CDK 4/6 Inhibitor
Brief Title: Study of Ribociclib With Everolimus + Exemestane in HR+ HER2- Locally Advanced/Metastatic Breast Cancer Post Progression on CDK 4/6 Inhibitor.
Acronym: TRINITI-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011XUS29
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Results first posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
Keywords: HR-positive; HER2-negative; Advanced breast cancer; LEE011; ribociclib; everolimus; Afinitor; exemestane; Aromasin; CDK; CDK4; CDK6; CDK4/6; CDK4/6 inhibitor; Phase I; Phase II; ER-positive; PR-positive; Postmenopausal; adult
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Everolimus; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort A (Experimental): Ribociclib (250 mg daily), everolimus (2.5 mg daily) and exemestane (25 mg daily) taken orally for 28 days. If no DLTs occurred, progressed to Cohort B
  Interventions: Drug: Ribociclib; Drug: Everolimus; Drug: Exemestane
- Cohort B (Experimental): Ribociclib (300 mg daily), everolimus (2.5 mg daily) and exemestane (25 mg daily) taken orally
  Interventions: Drug: Ribociclib; Drug: Everolimus; Drug: Exemestane
- Cohort C (Experimental): Ribociclib (200 mg daily), everolimus (5 mg daily) and exemestane (25 mg daily) taken orally
  Interventions: Drug: Ribociclib; Drug: Everolimus; Drug: Exemestane
- Group 1 (Experimental): Ribociclib (300 mg daily), everolimus (2.5 mg daily) and exemestane (25 mg daily) taken orally
  Interventions: Drug: Ribociclib; Drug: Everolimus; Drug: Exemestane
- Group 2 (Experimental): Ribociclib (200 mg daily), everolimus (5 mg daily) and exemestane (25 mg daily) taken orally
  Interventions: Drug: Ribociclib; Drug: Everolimus; Drug: Exemestane

INTERVENTIONS:
Drug: Ribociclib — supplied in 50 mg, 200 mg capsules/tablets taken orally and dosed daily for 28 day cycle
Drug: Everolimus — supplied in 2.5 mg tablets taken orally, daily for 28 day cycle
Drug: Exemestane — supplied in 25 mg tablets taken orally, daily for 28 day cycle

SUMMARY:
The purpose of this study is determine if the triplet combination of ribociclib, everolimus and exemastane is safe and effective in the treatment of locally advanced/metastatic breast cancer following treatment with a CDK 4/6 inhibitor

DETAILED DESCRIPTION:
This trial had two phases. The purpose of Phase I dose escalation and dose de-escalation was to determine the maximum tolerated doses (MTDs) and/or identify the recommended Phase II dose (RP2D) of the combination treatment of ribociclib+ everolimus + exemestane. The dosing was continuous in adult men and postmenopausal women with HR+ HER2-negative advanced breast cancer which was resistant to the non-steroidal aromatase inhibitors, fulvestrant or tamoxifen.

The purpose of the phase II portion of this trial was to evaluate the anti-tumor activity of exemestane, everolimus and ribociclib combination therapy following progression on a CDK 4/6 inhibitor.

The planned duration of the study was 30 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women
* Patient has a confirmed diagnosis of estrogen-receptor positive and/or progesterone receptor positive breast cancer by local laboratory and has HER2-negative breast cancer
* Patient must have either measurable disease by RECIST 1.1 or bone lesions in absence of measurable disease.
* ECOG Performance Status 0 - 1
* Disease refractory to either, AI, tamoxifen or fulvestrant
* Previously treated on any CDK 4/6 inhibitor.
* Patient has adequate bone marrow and organ function.

Exclusion Criteria:

* Patient with symptomatic visceral disease or any disease burden that makes the patient ineligible for endocrine therapy per the investigator's best judgment.
* Patient has received more than one line of chemotherapy for advanced disease.
* Previous treatment with mTOR inhibitors, or exemestane for advanced disease.
* Progressed on more than one CDK 4/6 inhibitor
* Patient with CNS involvement unless they are at least 4 weeks from prior therapy completion.
* Clinically significant, uncontrolled heart disease and/or recent cardiac events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Ironwood Cancer and Research Centers Ironwood Cancer, Chandler, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - UCLA Department of Medicine UCLA Hematology/Oncology, Los Angeles, California
  - University of California San Francisco Comprehensive Cancer Center, San Francisco, California
  - Central Coast Medical Oncology Corporation Onc Dept, Santa Maria, California
  - Yale University School of Medicine Smilow Cancer Hospital, New Haven, Connecticut
  - Florida Cancer Research Institute Dept of Oncology, Davie, Florida
  - Florida Cancer Specialists FL Cancer Specialists, Fort Myers, Florida
  - UF Health Cancer Center at Orlando Health UF Health (4), Orlando, Florida
  - Florida Cancer Specialists-North, St. Petersburg, Florida
  - Atlanta Cancer Center, Atlanta, Georgia
  - University of Kansas Cancer Center Univ of KS CC Medical Pavilion, Westwood, Kansas
  - Massachusetts General Hospital Mass Gen Hos Cancer Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - St. Luke's Cancer Institute Regulatory, Kansas City, Missouri
  - Research Medical Center HCA Midwest Division, Kansas City, Missouri
  - Washington University School of Medicine Washington U School of Medicin, St Louis, Missouri
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - University of Pennsylvania Medical Center Abramson Cancer Ctr of the Uni, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute Sarah Cannon Research Insti, Nashville, Tennessee
  - Oncology Consultants Oncology Consultants, Houston, Texas
  - MD Anderson Cancer Center/University of Texas MDACC, Houston, Texas
  - Huntsman Cancer Institute Huntsman Cancer Insti, Salt Lake City, Utah
  - Northwest Medical Specialties Dept of Onc, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  his trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cohort A, B and C were in Phase I and Group 1 and Group 2 classification were in Phase II
Period: Phase I
Arm/Group | Cohort A | Cohort B | Cohort C | Group 1 | Group 2
Started | 8 | 10 | 7 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 10 | 7 | 0 | 0
Not completed — Adverse Event | 1 | 3 | 1 | 0 | 0
Not completed — Progressive disease | 7 | 3 | 2 | 0 | 0
Not completed — Protocol deviation | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 3 | 4 | 0 | 0
Period: Phase II
Arm/Group | Cohort A | Cohort B | Cohort C | Group 1 | Group 2
Started | 0 | 0 | 0 | 46 | 33
Protocol Analysis Set (One patient had a major protocol deviation in Group II) | 0 | 0 | 0 | 46 | 32
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 46 | 33
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 3
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — Progressive dissease | 0 | 0 | 0 | 30 | 23
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 2 | 2
Not completed — Other | 0 | 0 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Cohort C | Group 1 | Group 2 | Total
Number analyzed (Participants) | 8 | 10 | 7 | 46 | 33 | 104
Age, Customized [Number; unit: participants]
  <40 years | 0 | 2 | 1 | 4 | 5 | 12
  ≥ 40 - < 50 years | 2 | 1 | 0 | 7 | 3 | 13
  ≥ 50 - < 60 years | 3 | 4 | 2 | 15 | 11 | 35
  ≥ 60 - < 70 years | 2 | 2 | 2 | 14 | 11 | 31
  ≥ 70 years | 1 | 1 | 2 | 6 | 3 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 7 | 46 | 33 | 104
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 1 | 1 | 2
  Black | 1 | 1 | 1 | 0 | 2 | 5
  White/Caucasian | 7 | 6 | 6 | 36 | 30 | 85
  Unknown | 0 | 2 | 0 | 5 | 0 | 7
  Other | 0 | 1 | 0 | 4 | 0 | 5
Body Mass Index [Number; unit: participants]
  < 30 BMI | 5 | 7 | 2 | 26 | 19 | 59
  ≥ 30 BMI | 3 | 3 | 4 | 18 | 11 | 39
  Missing | 0 | 0 | 1 | 2 | 3 | 6
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG: 0 - Fully active, able to carry on all pre-disease performance without restriction, 1 - Restricted in physically-strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  Participants
    Performance = 0 | 4 | 4 | 1 | 27 | 21 | 57
    Performance = 1 | 4 | 6 | 6 | 19 | 12 | 47

OUTCOME MEASURES:

1. Primary Outcome: Participants With Dose Limiting Toxicities by Preferred Term in Cycle 1 (28 Days) - in Phase I
Description: A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value assessed as having a reasonably possible relationship to the study medication(s) and is unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first 28 days of treatment (cycle 1) and meets any of the criteria defined in the protocol. National Cancer Institute Common Terminology Criteria for Adverse events (NCI CTCAE) version 4.03 will be used for all grading.
Time Frame: Baseline up to 28 days
Population: dose limiting toxicity-determining set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 8 | 10 | 7
Participants
  Febrile neutropenia Grade 3 | 1 | 1 | 0
  Neutropenia Grade 4 | 0 | 1 | 0
  Thrombocytopenia Grade 4 | 0 | 1 | 0
  Cardiac tamponade Grade 4 | 1 | 0 | 0
  Diarrhea Grade 3 | 1 | 0 | 0
  Hyperglycemia Grade 4 | 0 | 0 | 1

2. Primary Outcome: Clinical Benefit Rate as Per Central Review by Group- Phase II
Description: Clinical Benefit Rate (CBR) is defined as the percentage of participants with a complete response (CR) or partial response (PR) or with stable disease (SD) as per Response Evaluation Criteria in Solid Tumors (RECIST) V1.1 or Non-Complete Response or Non-Progressive Disease (NCRNPD) during first 24 weeks of first dose. CR=disappearance of all non-nodal target lesions, PR=at least a 30% decrease in the sum of diameter of all target lesions, SD=neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease (PD), PD=at least a 20% increase in the sum of diameter of all target lesions.
  The hypothesis was to be rejected if the lower limit of the 95% Confidence Interval for Clinical Benefit Rate (CBR) was greater than 10%.
Time Frame: From baseline up to 24 weeks
Population: Protocol analysis set. n: Number of patients who are at the corresponding category. ORR: percentage of patients having BOR of CR/PR.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 46 | 32
percentage of participants
  Overall response rate (CR+PR): | 6.5 [1.4 to 17.9] | 9.4 [2.0 to 25.0]
  CBR - CR+PR+SD (NCRNPD) by 24 weeks | 65.2 [49.8 to 78.6] | 59.4 [40.6 to 76.3]
  Disease control rate (CR+PR+SD(NCRNPD) | 65.2 [49.8 to 78.6] | 59.4 [40.6 to 76.3]

3. Primary Outcome: Best Overall Responses (BOR) Summary Table as Per Central Review by Group - Phase II
Description: Complete response (CR) or partial response (PR), or stable disease (SD) at 24 weeks as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or Non-CR Non-PD (NCRNPD) at Week 24.
Time Frame: Baseline up to 24 weeks and at 24 weeks
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 46 | 32
Participants
  Participants with measurable disease at baseline | 35 | 21
  Participants with non-measurable disease at baseline | 11 | 11
  Complete response (CR) | 0 | 0
  Partial Response (PR) | 3 | 3
  Stable disease (SD) | 17 | 6
  Progressive disease (PD) | 14 | 12
  NCRNPD - Non-complete response non-progressive disease | 10 | 10
  Unknown | 2 | 1

4. Secondary Outcome: Everolimus Pharmacokinetic Plasma Concentrations by Cohort - Phase I
Description: Plasma concentrations; below limit of quantitation values set to zero
Time Frame: Cycle 1,2: Day 1 and 15 - pre-dose, 2 and 4 hour post dose, Cycle 3 , Day 1 - pre-dose
Population: Pharmacokinetic analysis set. Number of participants with valid samples varied across timepoints and visits
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 8 | 10 | 7
ng/mL
  Cycle 1, Day 15 Pre-dose: number analyzed (Participants) | 3 | 6 | 7
  Cycle 1, Day 15 Pre-dose | 7.82 [3.57 to 10.3] | 8.31 [1.68 to 14.8] | 8.28 [5.25 to 15.0]
  Cycle 1, Day 15 2 H, post dose: number analyzed (Participants) | 3 | 5 | 7
  Cycle 1, Day 15 2 H, post dose | 15.2 [13.2 to 36.2] | 17 [6.84 to 34.4] | 36.2 [19.4 to 63.4]
  Cycle 1, Day 15 4 H, post dose: number analyzed (Participants) | 3 | 5 | 7
  Cycle 1, Day 15 4 H, post dose | 17.7 [16.7 to 18.5] | 16.2 [4.69 to 20.7] | 21.5 [13.6 to 35.8]
  Cycle 2, Day 1 Pre-dose: number analyzed (Participants) | 5 | 5 | 7
  Cycle 2, Day 1 Pre-dose | 6.47 [5.63 to 11.5] | 6.22 [1.71 to 10.5] | 7.76 [4.58 to 15.4]
  Cycle 2, Day 15 Pre-dose: number analyzed (Participants) | 5 | 6 | 5
  Cycle 2, Day 15 Pre-dose | 5.89 [4.33 to 9.52] | 4.26 [0.82 to 8.02] | 7.17 [5.4 to 15.3]
  Cycle 2, Day 15 2 H post-dose: number analyzed (Participants) | 4 | 5 | 6
  Cycle 2, Day 15 2 H post-dose | 21.8 [13.5 to 33.3] | 14.5 [8.67 to 30.1] | 22.1 [10.4 to 72.0]
  Cycle 2, Day 15 4 H post-dose: number analyzed (Participants) | 5 | 5 | 4
  Cycle 2, Day 15 4 H post-dose | 13.7 [5.42 to 20.7] | 9.13 [6.62 to 15.7] | 26.9 [20.5 to 41.1]
  Cycle 3, Day 1 4 H pre-dose: number analyzed (Participants) | 8 | 5 | 4
  Cycle 3, Day 1 4 H pre-dose | 4.7 [3.05 to 9.98] | 6.97 [2.87 to 22.5] | 6.33 [4.8 to 7.85]

5. Secondary Outcome: Best Overall Responses (BOR) Summary Table as Per Central Review by Cohort - Phase I
Description: Complete response (CR) or partial response (PR), or stable disease (SD)as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or Non-CR Non-PD (NCRNPD)
Time Frame: From baseline up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 8 | 10 | 7
Participants
  Participants with measurable disease at baseline | 5 | 7 | 4
  Participants with non-measurable disease at baseline | 3 | 3 | 3
  Complete response (CR) | 0 | 0 | 0
  Partial Response (PR) | 0 | 1 | 2
  Stable disease (SD) | 3 | 6 | 2
  Progressive disease (PD) | 3 | 0 | 0
  NCRNPD - Non-complete response non-progressive disease | 2 | 1 | 3
  Unknown | 0 | 2 | 0

6. Secondary Outcome: Clinical Benefit Rate as Per Central Review by Dose Cohort - Phase I
Description: Clinical Benefit Rate (CBR) is defined as the percentage of patients with a complete response (CR) or partial response (PR) or with stable disease (SD) at 24 weeks as per Response Evaluation Criteria in Solid Tumors (RECIST) V1.1 or Non-Complete Response Non-Progressive Disease (NCRNPD) up to Week 24 and at Week 24.
Time Frame: Baseline up to 24 weeks and at week 24
Population: Protocol analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 8 | 10 | 7
percentage of participants
  Overall response rate (CR+PR):: number analyzed (Participants) | 0 | 1 | 2
  Overall response rate (CR+PR): |  | 10.0 [0.3 to 44.5] | 28.6 [3.7 to 71.0]
  CBR - CR+PR+SD (NCRNPD) by 24 weeks: number analyzed (Participants) | 5 | 8 | 7
  CBR - CR+PR+SD (NCRNPD) by 24 weeks | 62.5 [24.5 to 91.5] | 80.0 [44.4 to 97.5] | 100.0 [59.0 to 100]
  CBR - CR+PR+SD (NCRNPD) at 24 weeks: number analyzed (Participants) | 5 | 8 | 7
  CBR - CR+PR+SD (NCRNPD) at 24 weeks | 0 [0.0 to 36.9] | 0.0 [0.0 to 30.8] | 28.6 [3.7 to 71.0]
  Disease control rate (CR+PR+SD(NCRNPD): number analyzed (Participants) | 5 | 8 | 7
  Disease control rate (CR+PR+SD(NCRNPD) | 62.5 [24.5 to 91.5] | 80.0 [44.4 to 97.5] | 100 [59.0 to 100]

7. Secondary Outcome: Summary of Progression-free Survival (PFS) (Months), as Per Central Review by Group - Phase II
Description: Progression is defined as <= 12 weeks after randomization/ start of treatment (and not qualifying for CR, PR or SD).
Time Frame: Baseline up to approximately 32 months
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 46 | 32
months | 8.0 [3.8 to 14.5] | 4.7 [2.0 to 12.7]

8. Secondary Outcome: Overall Survival (OS) by Group - Phase II
Description: Overall survival is the time from date of first treatment to the date of death due to any cause. If a patient is not known to have died, survival will be censored at the last date of contact.
Time Frame: Baseline up to approximately 32 months
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 46 | 32
months | 27.4 [16.8 to NA] — Not estimable - insufficient number of participants with events | NA [16.4 to NA] — Not estimable - insufficient number of participants with events

9. Secondary Outcome: Duration of Overall Response (DOR) by Group - Phase II
Description: Patients whose best response is complete response (CR) or partial response (PR). The start date is the date of first documented response (CR or PR) and the end date is the date of first documented progression or death due to underlying cancer.
Time Frame: Baseline up to approximately 16 months
Population: Full analysis set. N=number patients included in the analysis (with confirmed CR or PR)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 3 | 3
months | 14.6 [NA to NA] — Not estimable - insufficient number of participants with confirmed response to calculate CI upper and lower limits | 6.4 [5.5 to 7.4]

10. Secondary Outcome: Time to Definitive Deterioration of ECOG Performance Status in One Category of the Score by Group - Phase II
Description: Time to definitive deterioration of ECOG performance status in one category of score is defined as the time from the date of randomization to the date of event, which is defined as at least one score lower than the baseline.
Time Frame: Baseline up to approximately 8 months
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: median
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 46 | 32
median | NA [7.4 to NA] — Not estimable - insufficient number of participants with events | 12.0 [7.3 to NA] — Not estimable - insufficient number of participants with events

11. Secondary Outcome: Everolimus Pharmacokinetic Plasma Concentrations - Phase II
Description: Plasma concentrations; below limit of quantitation values set to zero
Time Frame: Cycle 1,2: Day 1 and 15 - pre-dose, 2 and 4 hour post dose, Cycle 3 , Day 1 - pre-dose
Population: Pharmacokinetic analysis set. Number of participants with valid samples varied across timepoints and visits
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 46 | 33
ng/mL
  Cycle 1, Day 15 pre dose: number analyzed (Participants) | 45 | 30
  Cycle 1, Day 15 pre dose | 214 [13.8 to 1410] | 132 [45.2 to 296]
  Cycle 1, Day 15 2 H post-dose: number analyzed (Participants) | 39 | 23
  Cycle 1, Day 15 2 H post-dose | 644 [38.6 to 2490] | 372 [83.8 to 686]
  Cycle 1, Day 15 4 H post-dose: number analyzed (Participants) | 39 | 23
  Cycle 1, Day 15 4 H post-dose | 583 [34.3 to 2320] | 323 [81.3 to 631]
  Cycle 2 Day 1 pre-dose: number analyzed (Participants) | 41 | 30
  Cycle 2 Day 1 pre-dose | 199 [2.27 to 691] | 125 [1.4 to 379]
  Cycle 2, Day 15 pre-dose: number analyzed (Participants) | 41 | 28
  Cycle 2, Day 15 pre-dose | 245 [21.2 to 1350] | 170 [2.72 to 382]
  Cycle 2, Day 15 2 H post-dose: number analyzed (Participants) | 36 | 24
  Cycle 2, Day 15 2 H post-dose | 652 [140 to 2260] | 442 [2.34 to 1240]
  Cycle 2, Day 15 4 H post-dose: number analyzed (Participants) | 37 | 24
  Cycle 2, Day 15 4 H post-dose | 642 [133 to 2130] | 406 [2.1 to 1040]
  Cycle 3, Day 1 pre-dose: number analyzed (Participants) | 26 | 20
  Cycle 3, Day 1 pre-dose | 193 [1.52 to 1080] | 198 [2.61 to 504]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 108 weeks
Groups:
- Cohort C: Ribociclib (200 mg daily), everolimus (5 mg daily) and exemestane (25 mg daily) taken ora
Arm/Group | Cohort A | Cohort B | Cohort C | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 6/8 | 5/10 | 0/7 | 20/46 | 11/33
Serious Adverse Events (participants affected / at risk) | 3/8 | 3/10 | 5/7 | 11/46 | 5/33
Other Adverse Events (participants affected / at risk) | 8/8 | 10/10 | 7/7 | 46/46 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=8) | Cohort B (N=10) | Cohort C (N=7) | Group 1 (N=46) | Group 2 (N=33)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1 | 3 | 2
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=8) | Cohort B (N=10) | Cohort C (N=7) | Group 1 (N=46) | Group 2 (N=33)
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 6 | 12 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 2 | 4 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 7 | 5 | 20 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2 | 2 | 15 | 8
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 3 | 2
Eye oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 4 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1 | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 4
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 2 | 17 | 8
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 3 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 5 | 1
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 5 | 0 | 17 | 11
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 4 | 3 | 24 | 11
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 6 | 7
Asthenia (General disorders) | 0 | 1 | 0 | 1 | 0
Axillary pain (General disorders) | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 4 | 3
Fatigue (General disorders) | 4 | 2 | 5 | 19 | 10
Influenza like illness (General disorders) | 0 | 1 | 0 | 2 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 3
Non-cardiac chest pain (General disorders) | 0 | 2 | 0 | 2 | 3
Oedema peripheral (General disorders) | 1 | 0 | 6 | 10 | 8
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 10 | 5
Seasonal allergy (Immune system disorders) | 0 | 2 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 3 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Groin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 1 | 1
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Nail bed infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 2 | 2
Onychomycosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 3 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 6 | 3
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 2 | 8 | 4
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 8 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Alanine aminotransferase decreased (Investigations) | 0 | 0 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 8 | 5
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase decreased (Investigations) | 0 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 3 | 12 | 7
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 3 | 4 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 2 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 3 | 4 | 1
Blood folate decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 3 | 1
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 3 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 3 | 5 | 4
High density lipoprotein decreased (Investigations) | 0 | 0 | 1 | 0 | 0
High density lipoprotein increased (Investigations) | 0 | 0 | 1 | 0 | 0
Lipase decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 2 | 0 | 1 | 1 | 2
Low density lipoprotein increased (Investigations) | 0 | 0 | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 1 | 2 | 16 | 10
Platelet count decreased (Investigations) | 1 | 1 | 0 | 5 | 4
Platelet count increased (Investigations) | 0 | 0 | 1 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 2 | 1 | 2 | 6 | 4
White blood cell count decreased (Investigations) | 2 | 3 | 2 | 13 | 6
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 6 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 3 | 6 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 4 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 5 | 9 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 5 | 8 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 13 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 9 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 5 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 5 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 4
Dysgeusia (Nervous system disorders) | 1 | 1 | 1 | 11 | 4
Headache (Nervous system disorders) | 1 | 1 | 1 | 7 | 9
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 4 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 2 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1 | 3
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 7 | 5
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 3
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 3 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 10 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 5 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 6 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 3
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 7 | 4
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 5 | 5 | 8 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 4 | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0 | 6 | 3
Hypertension (Vascular disorders) | 0 | 1 | 1 | 4 | 2
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 1 | 1 | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT02732119/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT02732119/SAP_001.pdf